CLINICAL TRIAL: NCT00003966
Title: Defibrotide for Hematopoietic Stem Cell Transplant Patients With Severe Hepatic Venocclusive Disease: A Phase I/II Study to Determine the Minimal Effective Dose
Brief Title: Defibrotide in Treating Patients With Liver Damage Following Peripheral Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Jazz Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul G. Richardson, MD, Richardson, Paul MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99118; P30CA015704 (NIH); DFCI-1999-P-010076/14; DUMC-00176-00-2; FHCRC-1375.00; NCI-G99-1548; CHNMC-02118; MSKCC-03-058; JHMI-00-06-02-02
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Veno-occlusive Disease
Keywords: veno-occlusive disease
MeSH Terms: interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A Lower dose (Experimental): This is a randomized, multicenter study. All patients initially receive the same dose of defibrotide IV over 2 hours every 6 hours on day 1. On day 2, patients are randomized to 1 of 2 doses of defibrotide.
  - Arm I: On days 2-14, patients receive a lower dose of defibrotide IV over 2 hours every 6 hours.
  In both arms, courses repeat every 14 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: defibrotide
- Arm B Higher Dose (Experimental): This is a randomized, multicenter study. All patients initially receive the same dose of defibrotide IV over 2 hours every 6 hours on day 1. On day 2, patients are randomized to 1 of 2 doses of defibrotide.
  - Arm II: On days 2-14, patients receive a higher dose of defibrotide IV over 2 hours every 6 hours.
  In both arms, courses repeat every 14 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: defibrotide

INTERVENTIONS:
Drug: defibrotide
  Other Names: Defitelio®

SUMMARY:
RATIONALE: Giving defibrotide may be an effective treatment for liver damage that may result following peripheral stem cell transplantation.

PURPOSE: This randomized phase II trial is studying defibrotide to see how well it works in treating patients with severe liver disease after undergoing peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine complete response rate in post-hematopoietic stem cell transplant patients with severe veno-occlusive disease of the liver treated with defibrotide.
* Determine the minimal effective dose of this drug in these patients.
* Assess toxicity and adverse side effects of this drug in these patients.

OUTLINE: This is a randomized, multicenter study. All patients initially receive the same dose of defibrotide IV over 2 hours every 6 hours on day 1. On day 2, patients are randomized to 1 of 2 doses of defibrotide.

* Arm I: On days 2-14, patients receive a lower dose of defibrotide IV over 2 hours every 6 hours.
* Arm II: On days 2-14, patients receive a higher dose of defibrotide IV over 2 hours every 6 hours.

In both arms, courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 140 patients (70 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of VOD defined by:

  * Jaundice (bilirubin ≥ 2 mg/dL) and 2 or more of the following: ascites, weight gain > 5% above baseline weight (see Section 5.2), hepatomegaly, RUQ pain

    * Patients with jaundice and reversal of flow on Doppler examination of the portal vein will be eligible with one of the following: ascites, weight gain > 5% above baseline weight, hepatomegaly, RUQ pain
    * Patients with pre-existing hepatomegaly must have documentation by physical exam or imaging that liver size is increased over baseline at admission
  * Patients who do not meet the criteria in Section 3.1.1 (ie. have two of the major criteria but not three) and have biopsy proven VOD are eligible in the presence of characteristics consistent with severe disease (see below).
  * Patients with concurrent, confounding causes of liver dysfunction clinically evident or evident on ultrasound or other radiographic imaging (such as evidence of biliary ductal dilatation or focal tissue defects) may require biopsy-proven VOD and/or elevated wedged trans-hepatic venous pressure gradient measurement ( ≥10 mm mercury) to be considered eligible. Best medical judgment and further imaging studies can be used to clarify the diagnosis and determine confounding causes of liver dysfunction.
* Severity of VOD defined by:

  * For patients addressed by the Bearman model (i.e. within 16 days of SCT and conditioned with either BU/CY, CY/TBI or CBV), there must be a 30% or greater risk of severe VOD (see Appendix B).
  * For all other patients who are not addressed by the Bearman model (ie. beyond 16 days of SCT and/or not conditioned with either BU/CY,
  * CY/TBI or CBV), there must be concomitant multi-organ failure defined as presence of one or more of the following :

    * renal dysfunction: a) creatinine ≥2x value on the date of admission day to the BMT unit for conditioning or ≥2x lowest value during conditioning (use the lowest value for calculation), or b) creatinine clearance or GFR ≤50% of admission value, or c) dialysis dependence"
    * pulmonary dysfunction: documentation of oxygenation saturation ≤ 90% on room air; requirement for positive pressure/ventilator dependence

      ----pulmonary dysfunction must not be attributable to another cause (e.g. documented infectious pneumonia)
    * central nervous dysfunction: documentation of confusion, lethargy, and/or delirium ---- central nervous dysfunction must not be attributable to another cause (e.g. documented cyclosporin toxicity)
  * Patients or their parents/guardians or designated proxy must have the ability to give voluntary informed consent to the protocol. Where possible, patient assent will also be obtained
  * Patients must be ≥ 12 hours after cessation of heparin
  * Patient must have an eligible diagnosis of VOD by Day 35 post transplant
* Exclusion Criteria

  * Patients receiving concomitant heparin or other anticoagulants unless being used for routine CVL management, fibrinolytic instillation for CVL occlusion, intermittent dialysis or ultrafiltration are excluded. Patients who have received systemic t-PA (concomitant or prior) are excluded.
  * Patients with significant uncontrolled acute bleeding, defined as hemorrhage requiring > 15 cc/kg of packed red blood cells (ie. a pediatric patient weighing 20 kg and requiring > 300cc of packed red blood cells /24 hours or an adult patient weighing 70 kg and requiring >3 units of packed red blood cells/24 hours) to replace blood loss are excluded. These parameters must be reviewed prior to enrollment by the PI or his/her designate.
  * Patients with hemodynamic instability as defined below:

    * Hemodynamic stability is defined as having no requirement for pressor support OR being able to maintain mean arterial pressure within 1 SD of age-adjusted levels with pressor support (see Appendix D)
    * Patients requiring renal dose dopamine alone (2-5 mcg/kg/min) are eligible without measurement of mean arterial pressure
  * Patients with Grade B-D GVHD, graded according to the IBMTR Severity Index (see Appendix G). Please note patients with Grade B skin only are eligible.
  * Patients intubated for documented intrinsic lung disease

    --- Patients intubated secondary to a mechanical barrier to ventilation, e.g.pulmonary edema or ascites, will be eligible as long as the PaO2/FiO2 ratio is ≥ 300 and/or the oxygen index (OI={MAP x FiO2}÷ PaO2 x 100) is ≤ 25% at the time of enrollment
  * Patients who meet Grade IV common toxicity criteria for neurotoxicity (other than Grade IV confusion and/or delirium), i.e. coma, seizures, toxic psychosis
  * Patients who are currently receiving treatment with another experimental agent.
  * Please note that an experimental agent in this setting is defined as any drug or device used under an IND designation which is associated with systemic effects that could influence the outcome in a patient with severe VOD. If the continued use of an experimental agent is considered both necessary and appropriate, this must be reviewed and approved on a case by case basis by the Overall Study PI, Dr. Paul Richardson, or his designate, who will approve the entry of patients being concurrently treated with another experimental agent only if there is no evidence for a potential adverse pharmacokinetic interaction or overlapping toxicity.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2000-04; Primary Completion 2006-02 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate as measured by a total bilirubin of < 2 mg/dL and resolution of multi-organ failure attributable to veno-occlusive disease (VOD) | 60 Days

SECONDARY OUTCOMES:
Survival at 100 days following stem cell transplantation | 100 days following stem cell transplantation
Toxicity by NCI Common Toxicity Criteria version 2.0 during study and 30 days after study completion | during study and 30 Days after study completion
Grade 3-4 end organ dysfunction attributable to defibrotide as determined by NCI Common Toxicity Criteria version 2.0 during study and 30 days after study completion | during study and 30 Days after study completion
Occurrence of other adverse events by NCI Common Toxicity Criteria version 2.0 during study and 30 days after study completion | during study and 30 Days after study completion
Effect of drug on plasminogen activator inhibitor-1 (PAI-1) determination of dose-relationship between drug and/or VOD response as measured by survival, PAI-1 levels, and research assays at day 100 | 100 Days
Feasibility of pharmacokinetics (PK) across dose arms and the PK of defibrotide by PK analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Richardson PG, Soiffer RJ, Antin JH, et al.: Defibrotide (DF) for the treatment of severe veno-occlusive disease (VOD) and multi-system organ failure (MOF) post SCT: final results of a phase II, multicenter, randomized study and preliminary analyses of surrogate markers and ultrasound findings. [Abstract] Blood 104 (11): A-350, 2004.
- [Result] Richardson P, Soiffer RJ, Antin JH, et al.: Defibrotide (DF) is effective in the treatment of severe veno-occlusive disease (VOD) and multi-system organ failure (MOF) post stem cell transplantation (SCT): results of a phase II, multicenter, randomized study. [Abstract] Blood 102 (11): A-674, 2003.
- [Result] Richardson PG, Soiffer R, Antin JH, et al.: Defibrotide (DF) appears effective and safe in a phase II, randomized study of patients (pts) with severe veno-occlusive disease (VOD) and multi-system organ failure (MOF) post stem cell transplantation (SCT). [Abstract] Blood 100 (9): A-414, 2002.